CLINICAL TRIAL: NCT00769093
Title: Pilot Study to Compare Dynamic MR Imaging Changes in Patients With Recurrent High Grade Glioma, Receiving an Antiangiogenic Drug, Bevacizumab, Versus Dexamethasone. Dual Agent MR Imaging Study, Using Gadolinium and Ferumoxytol (Code 7228)
Brief Title: Assessing Dynamic Magnetic Resonance (MR) Imaging in Patients With Recurrent High Grade Glioma Receiving Chemotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Edward Neuwelt, Professor, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00003678; 26XS293 (Other Grant/Funding Number: NCI SAIC-Frederick Contract); 3678 (Other: OHSU eIRB); SOL-07083-LX (Other: OHSU Knight Cancer Institute); OHSU-3678 (Other: OHSU IRB)
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Brain Neoplasms
Keywords: ferumoxytol; diagnostic imaging
MeSH Terms: conditions — Brain Neoplasms | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Both groups will receive an intravenous chemotherapeutic drug (carboplatin). The first study group (n=6) will receive bevacizumab, the antiangiogenic agent for three weeks, then dexamethasone for three weeks.
  Interventions: Drug: Ferumoxytol
- Group 2 (Active Comparator): Both groups will receive an intravenous chemotherapeutic drug (carboplatin). The second study group (n=6) will receive dexamethasone for 3 weeks, then switch to bevacizumab, the antiangiogenic agent, for 3 weeks.
  Interventions: Drug: Ferumoxytol

INTERVENTIONS:
Drug: Ferumoxytol — 2 mg/kg
  Other Names: AMAG Pharmaceuticals, Inc., Code 7228

SUMMARY:
The purpose of this study is to learn more about imaging changes induced by a new therapeutic agent, bevacizumab with the standard steroid, dexamethasone in patients with high grade glioma. Magnetic resonance imaging (MRI) will be used to evaluate the difference between the 2 treatments. The usual contrast agent (gadolinium) and an iron containing contrast agent called "ferumoxytol" may help us to evaluate the differences between bevacizumab and dexamethasone effects on imaging of a brain tumor called high grade glioma. For this purpose, after intravenous contrast agent injection, special MR scans (called: dynamic perfusion, blood-brain barrier (BBB) permeability measurement) will be performed to see the microvascular changes in the brain and tumor.

DETAILED DESCRIPTION:
Adult patients (>18 years old) with recurrent high grade glioma (confirmed by radiology and tissue sample), who have progressed on prior temozolomide + radiation therapy, will be recruited from the neurology, neurosurgery, or neuro-oncology clinics. Patients will be enrolled if they meet the study inclusion and exclusion criteria

Patients will be scanned at four different time-points (4 MRI series) (1) before the beginning of the treatment (base line), (2) Three weeks after the first treatment, (3) Three weeks after the second treatment, and (4) at time of progression of the disease. Each MRI time-point will consist of a series of MRI's on three consecutive days. On the first day, gadolinium (0.1 mmol/kg) will be injected for the MRI scan. On the following day ferumoxytol (2 mg/kg) and on the third day, the MRI scan will be done without additional contrast agent, to see the delayed contrast enhancement of ferumoxytol.

Subjects will be on treatment including a chemotherapeutic agent called carboplatin combined with either bevacizumab or dexamethasone; 6 patients will receive carboplatin-bevacizumab, followed by carboplatin-dexamethasone, another 6 patients will receive carboplatin- dexamethasone, followed by carboplatin-bevacizumab. After the 3rd time-point, all the patients will continue on carboplatin-bevacizumab treatment (which is currently not an FDA approved combination for brain tumors, however it is widely used throughout the country).There will be monthly clinical visits with clinical MRI until progression of the disease. There will be a follow up visit, 1 month after the last ferumoxytol injection.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age equal or greater than 18 years
* Histologically confirmed high grade glioma
* Radiographic demonstration of disease progression following prior therapy of temozolomide + radiation
* Patient scheduled for bevacizumab + standard IV chemotherapy therapy
* Bi-dimensionally measurable disease on gadolinium enhanced T1 weighted MR scans
* An interval of at least 4 weeks since prior surgical resection
* Patients corticosteroid dose must be 4 mg per day or less.
* Karnofsky performance status greater than or equal to 50
* Life expectancy greater than 12 weeks
* Ability to comply with study and follow-up procedures

Exclusion Criteria:

* Pregnant or nursing females
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known liver function insufficiency, stage IV or V renal insufficiency
* Disease and Treatment History: Prior treatment with bevacizumab, or another vascular endothelial growth factor (VEGF) or VEGFR-targeted agent; Need for urgent palliative intervention for primary disease (e.g., impending herniation
* Bevacizumab Exclusion Criteria: History of hypertensive encephalopathy; New York Heart Association (NYHA) Grade II or greater congestive heart failure (CHF); History of myocardial infarction or unstable angina within 6 months prior to start of the study; History of stroke or transient ischemic attack within 6 months prior to study enrollment; Significant vascular disease (e.g., aortic aneurysm, aortic dissection) or recent peripheral arterial thrombosis within 6 months prior to start of the study; Evidence of bleeding diathesis or coagulopathy; on therapeutic anti-coagulants.
* Subjects unable to undergo an MRI with contrast
* Ferumoxytol Exclusion Criteria: History of allergic reactions attributed to compounds of similar chemical or biologic composition to ferumoxytol: parenteral iron, parenteral dextran, parenteral iron-dextran, or parenteral iron-polysaccharide preparations (Ferumoxytol Investigator's Drug Brochure, 2005). Patients with significant drug or other allergies or autoimmune diseases may be enrolled at the Investigator's discretion
* Subjects with known or suspected iron overload (genetic hemochromatosis or history of multiple transfusions).Patients with transferrin saturation greater than 60%
* Inability or unwillingness to undergo the complete series of imaging sessions. Inability or unwillingness to return to the neuro-oncology clinic at Oregon Health and Science University (OHSU) for the one month follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The primary objective of this project is to describe quantitative imaging changes of brain tumor vascularity after anti-angiogenic therapy versus steroid therapy. This objective will be accomplished with the following aims and associated hypotheses. | 15 weeks
To describe changes of quantitative blood brain barrier permeability measurements (Ktrans) of a standard gadolinium (Gd) MRI contrast between bevacizumab anti-angiogenic therapy and dexamethasone. | 15 weeks
To describe relative cerebral blood volume (rCBV) changes obtained using ferumoxytol an iron oxide nanoparticle blood pool agent. | 15 weeks

SECONDARY OUTCOMES:
To assess vascular dynamic parameters (rCBV and Ktrans) values at progression. | at progression
To describe the changes of the vascular dynamic parameters (rCBV, Ktrans) with the changes of standard gadolinium enhancing tumor volume | 15 weeks
To describe post contrast tumor volume (enhancement) of gadolinium and ferumoxytol. | 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Neuwelt, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States